CLINICAL TRIAL: NCT06456762
Title: Developing and Testing a Text-messaging Intervention to Support Parents After Their Child's Psychiatric Emergency
Brief Title: Text-messaging Intervention to Support Parents After Their Child's Psychiatric Emergency
Acronym: iPEACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Margaret M. Benningfield, Associate Professor of Psychiatry and Behavioral Sciences, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 231812; R34MH132711-01A1 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Parents; Self Efficacy; Mental Health Literacy; Psychiatric Emergency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iPEACE: Intervention for Parent Education About Care after the ED (Active Comparator): Parents in the iPEACE condition will receive an 8-week text-messaging intervention to build skills in mental health literacy and self-efficacy. Texts will be delivered several days per week over an 8-week period. The intervention is fully automated.
  Interventions: Behavioral: iPEACE: Intervention for Parent Education about Care after the ED
- Text Reminders Only (Active Comparator): Parents in the text-reminders only condition will receive weekly reminders to make an outpatient therapy appointment for their child. Texts will be fully automated, and will be delivered once a week for 8-weeks.
  Interventions: Behavioral: Text Messaging Reminders Only
- Treatment as Usual (No Intervention): Parents in the TAU condition will receive typical treatment in the emergency department, including outpatient referrals and safety planning if needed prior to discharge.

INTERVENTIONS:
Behavioral: iPEACE: Intervention for Parent Education about Care after the ED — Automated texting intervention for parents to increase engagement in their child's outpatient mental health treatment over an 8-week period.
  Arms: iPEACE: Intervention for Parent Education About Care after the ED
Behavioral: Text Messaging Reminders Only — Weekly automated text reminders to instruct parents to make an appointment with their child's outpatient mental health provider over an 8-week period.
  Arms: Text Reminders Only

SUMMARY:
This grant aims to develop and test a text-messaging intervention for parents of children and teens evaluated in the emergency department for a psychiatric emergency and discharged home with outpatient referrals. The intervention for parents will teach parents skills to navigate the mental health services system and build their self-efficacy in managing their child's mental health. This research has the potential to improve services for families seeking emergency psychiatric support, with the goal of facilitating treatment engagement and reducing emergency services utilization using scalable, cost-effective, accessible tools.

DETAILED DESCRIPTION:
Rates of emergency department (ED) visits for psychiatric emergencies in adolescents have increased substantially in the past decade, including for suicidality, self-harm, and aggression. A substantial number of these adolescents will be discharged home from the ED with referrals to outpatient mental health treatment. Yet, engagement in outpatient mental health treatment among adolescents is low, and rates of repeated emergency services utilization are high, highlighting the need for better supports for these youth and families. While effective, brief interventions have been developed to directly support adolescents at the time of their ED visit, no evidence-based interventions have been developed to support parents of these youth. Further, the period following an emergency visit is known to be high risk, yet no existing services support parents during the transition home, while waiting for connection to outpatient services. In this intervention development study, the investigators seek to iteratively develop, refine, and test an automated, text-messaging intervention for parents of youth discharged from the ED after a psychiatric emergency. The 8-week intervention (iPEACE; intervention for parent education after care in the ED) will directly target (1) parent mental health literacy and (2) parent self-efficacy, with the goal of reducing ED utilization and enhancing outpatient mental health service use and engagement. In the first phase of the study, the investigators aim to develop and refine the intervention with stakeholder feedback. Parents (N=15) will receive the 8-week iPEACE starting immediately following ED discharge. Parents will provide both in-the-moment feedback via text-message surveys and in-depth feedback at the end of the 8-week period via semi-structured qualitative interviews and self-report measures. The investigators will also conduct qualitative interviews with enrolled parents' children and key ED stakeholders. The investigators will use this feedback to refine the intervention materials. In the second phase of the study, the investigators will conduct a pilot randomized controlled trial (N=90), with n=30 parents randomized to enhanced usual care, n=30 randomized to enhanced usual care with text-message reminders, and n=30 randomized to receive iPEACE. Parents and their child evaluated in the ED will complete follow-up assessments at 4-, 8- and 24-weeks to assess key intervention targets (self-efficacy and mental health literacy) and youth outcomes (outpatient mental health service utilization, ED utilization, clinical symptom severity). The goals for the proposed project include: (1) developing and refining the iPEACE text-messaging intervention; and (2) piloting the iPEACE intervention compared to enhanced usual care only and enhanced usual care with text-message reminders to assess key study outcomes and mechanisms to inform a fully-power randomized trial. This R34 has important clinical implications, as findings from this study may support the testing and implementation of a digital health intervention to improve outcomes for high-risk youth and families. The proposed study has the potential to inform the provision of clinical services to support families during high-risk clinical transitions.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardians of a child ages 11-17;
* Parents or legal guardians must live with their child ≥50% of the time;
* Child must be admitted to the pediatric emergency department for a mental health crisis;
* Child must be discharged home from the emergency department with referrals to outpatient care.

Exclusion Criteria:

* Do not have daily access to a mobile phone that can receive SMS text messages;
* Do not speak and read fluently in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Services Assessment: Outpatient Mental Health Service Utilization | 24 weeks
  The Child and Adolescent Services Assessment will be used as a parent self-report measure that evaluates the total number of outpatient mental health appointments the participant's child attends during the follow-up period. The outcome will be a total count of the number of outpatient mental health appointments attended.
Child and Adolescent Services Assessment: Emergency Department Services Use | 24 weeks
  The Child and Adolescent Services Assessment will be used as a parent self-report measure to evaluate the number of psychiatric emergency department visits the participant's child has during the follow-up period. The outcome variable will be a dichotomous variable based on whether the child was readmitted to the emergency department during the follow-up period (yes/no).

SECONDARY OUTCOMES:
Suicidal Ideation Questionnaire - Jr. | 24 weeks
  Child suicidal thoughts will be assessed using the Suicidal Ideation Questionnaire-Jr. child self-report measure over follow up period. Scores range from 0-90, with higher scores reflecting higher suicidal ideation severity. The clinical cutoff score is 31.
Self-Injurious Thoughts and Behaviors Interview - Revised | 24 weeks.
  Child suicidal thoughts and behaviors will be assessed using an adapted version of the Self-Injurious Thoughts and Behaviors Interview-Revised (SITBI-R); the study will use a child self-report version of the SITBI-R. The SITBI-R will provide outcome scores on the presence or absence of a suicide attempt during the follow up period and the presence or absence of passive and active suicidal ideation during the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Benningfield, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share data in accordance with the National Institutes of Health data sharing policy. Researchers can use the standard request process through the NIMH Data Archive to request access to the research data. The NIMH Data Archive Data Access Committee makes decisions about granting research access, which is allowable for one year with an option to renew.Data provided to the NDA will be de-identified and all participants will consent to data sharing at the time of study enrollment. The NIMH Data Archive GUID allows researchers to aggregate data from a single research participant such that they remain deidentified.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will submit individual participant data to the NIMH NDA every 6-months for the duration of the study. Uploads of all scientific and meta-data will be harmonized, validated, and submitted at 6-month intervals over the course of the award, following standard January 15 and July 15th deadlines.